CLINICAL TRIAL: NCT05924919
Title: The Effects of Passive Heat Therapy in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20024906; 22-01741 (Other Grant/Funding Number: American College of Sports Medicine)
Record Dates: First submitted 2023-05-25; First posted 2023-06-29 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm: Whole-body Passive Heat Therapy (HT) (Experimental): Heat therapy will be administered using an infrared sauna. The intervention duration will last 25 minutes at a temperature of 60°C.
  Interventions: Procedure: Whole-body Passive Heat Therapy (HT); Procedure: Thermoneutral Control (CON)

INTERVENTIONS:
Procedure: Whole-body Passive Heat Therapy (HT) — The whole-body passive heat therapy (HT) intervention will consist of an acute bout of infrared sauna for 25 minutes at 60°C. Participants will lie supine on a memory foam pad.
Procedure: Thermoneutral Control (CON) — Participants will remain in a room temperature environment (22°C) underneath the infrared domes for 25 minutes.

SUMMARY:
The objective of this proposal is to investigate the acute effects of whole-body passive heat therapy using far-infrared technology on vascular function, exercise capacity, and renal function in CKD patients. The central hypothesis is that an acute bout of whole-body passive heat therapy will be well-tolerated and lead to acute improvements in large blood vessel (macrovascular) function, small blood vessel (microvascular) function, and exercise capacity without significantly altering markers of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria for participants with CKD:

* Age > 18 years old
* Stage 2-4 CKD

Exclusion Criteria for participants with CKD:

* Unstable medical conditions characterized by frequent or unpredictable biological, chemical, or psychological changes
* Uncontrolled hypertension
* Current fluid restrictions
* End stage kidney disease or currently on dialysis treatment
* Body weight < 40kg
* Exhibits any contraindications to exercise as per ACSM guidelines
* Regular tobacco and/or nicotine use
* History of heat-related illness
* Participates in regular exercise and/or sauna use
* Current hormone replacement therapy
* Pacemaker or electro-medical implant
* Persons with or at risk of intestinal disorders including gastroporesis
* History of diverticula
* Persons who have undergone surgical procedures in the GI tract
* Swallowing disorders
* Chron's disease
* Current pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Renal Safety of Heat Therapy | Change from baseline to 90 minutes after intervention
  Change in urinary NGAL
Tolerability of Heat Therapy as Assessed using Validated Questionnaires of Thermal Perception | During 25 minute intervention
  Self reported perception of heat using the the Thermal Sensation Scale.

SECONDARY OUTCOMES:
Conduit artery endothelial function | 90 minutes after intervention
  Brachial artery flow-mediated dilation assessed by high-resolution duplex ultrasound.
Lower Limb Microvascular Function | 90 minutes after intervention
  Lower limb microvascular function will be assessed with high-resolution duplex ultrasound during passive leg movement (PLM) technique.
Exercise Capacity | 90 minutes after intervention
  The 6-minute walk test distance.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kirkman, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No